CLINICAL TRIAL: NCT01796379
Title: High Intensity Training in de Novo Heart Transplant Recipients in Scandinavia
Acronym: HITTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Norwegian Health Association (Other)
Responsible Party: Principal Investigator, Kari Nytrøen, Post doc, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9378
Record Dates: First submitted 2013-02-18; First posted 2013-02-21 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Heart Transplant Recipients; Physical Fitness
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (Experimental)
  Interventions: Behavioral: High Intensity Interval Training
- Moderate Training (Other): Regular exercise training offered as usual care to all heart transplant recipients.
  Interventions: Behavioral: Moderate Training

INTERVENTIONS:
Behavioral: High Intensity Interval Training — 9 months of high intensity interval based aerobic exercise (3 times/week)
  Arms: High Intensity Interval Training
Behavioral: Moderate Training
  Other Names: Regular exercise training offered to all heart transplant recipients (usual care)
  Arms: Moderate Training

SUMMARY:
Compared to end-stage heart failure, a patient's situation is usually greatly improved after a heart transplant (HTx), but the exercise capacity remains sub-normal, also long-term, ranging from 50 to 70% in most studies. While effective rehabilitation, including regular exercise, is considered an effective tool of improving health related quality of life (HRQoL) and prognosis of cardiac patients in general, the knowledge about and the effect of different rehabilitation programs among HTx recipients is limited. Exercise training is considered one of the most central parts in rehabilitation, but the mode of exercise used in different studies varies considerably. It is documented that high intensity interval training (HIT) has superior effects compared to training with moderate intensity in cardiac and heart failure patients. In contrast, HTx recipients have a denervated heart, and HIT had been considered unphysiological. However, the investigators have recently demonstrated highly beneficial effects on exercise capacity, muscle strength, body composition, reduced progression of cardiac allograft vasculopathy and HRQoL among long-term HTx recipients. In the present study the investigators want to test the hypothesis that systematic aerobic exercise with high intensity improve exercise capacity also in newly transplanted recipients, and secondarily that it gives favourable effects on the heart, peripheral circulation and a better HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable HTx recipients approximately 8-12 weeks after HTx.
* Age > 18 years, both sexes
* Received immunosuppressive therapy as per local protocol.
* Patient willing and capable of giving written informed consent for study participation and anticipated to be able to participate in the study for 9- 12 months.

Exclusion Criteria:

* Unstable condition or postoperative complications
* Recent severe rejection episodes
* Physical disabilities which prevent participation
* Other diseases or disabilities that contradict/refrain from exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Effect of exercise on peak oxygen uptake | Baseline to one year
  Change in ml/kg/min

SECONDARY OUTCOMES:
Effect of exercise on muscle strength | Baseline to one year
  Change measured in Newtonmeter and Joule
Effect of exercise on progression of coronary artery vasculopathy (CAV) | Baseline to one year
  Change measured by intravascular ultrasound; change in maximum intimal thickness, total atheroma volume, percent atheroma volume and virtual histology.
Effect of exercise on chronotropic responses | Baseline to one year
  Change in heart rate response, including changes in minimum and maximum heart rate and changes in chronotropic response index.
Effect of exercise on myocardial function | Baseline to one year
  Change in echocardiographic parametres such as stroke volume, cardiac index and ejection fraction.
Effect of exercise on endothelial function | Baseline to one year
  Change in endothelial function measured by flow mediated dilatation and EndoPat
Effect of exercise on biomarkers | Baseline to one year
  Neuroendocrine, inflammatory and immunological biomarkers.
Effect of exercise on health related quality of life | Baseline to one year
  Change measured on visual analogue scales and questionnaires
Effect of exercise on safety and tolerability | Baseline to 3 years follow-up
  Measured by number of serious adverse effects related to the intervention
Long-term effects of exercise | Baseline to 3 years follow-up
  Long-term effects will be measured by all outcomes listed above, including number of serious adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, Professor, Principal Investigator — Oslo Unversity Hospital
Locations (3):
- Copenhagen University Hospital, Copenhagen, Denmark
- Oslo University Hospital Rikshospitalet, Oslo, Norway
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Nytroen K, Rustad LA, Aukrust P, Ueland T, Hallen J, Holm I, Rolid K, Lekva T, Fiane AE, Amlie JP, Aakhus S, Gullestad L. High-intensity interval training improves peak oxygen uptake and muscular exercise capacity in heart transplant recipients. Am J Transplant. 2012 Nov;12(11):3134-42. doi: 10.1111/j.1600-6143.2012.04221.x. Epub 2012 Aug 17. PMID 22900793
- [Background] Nytroen K, Yardley M, Rolid K, Bjorkelund E, Karason K, Wigh JP, Dall CH, Arora S, Aakhus S, Lunde K, Solberg OG, Gustafsson F, Prescott EI, Gullestad L. Design and rationale of the HITTS randomized controlled trial: Effect of High-intensity Interval Training in de novo Heart Transplant Recipients in Scandinavia. Am Heart J. 2016 Feb;172:96-105. doi: 10.1016/j.ahj.2015.10.011. Epub 2015 Oct 21. PMID 26856221
- [Background] Rolid K, Andreassen AK, Yardley M, Bjorkelund E, Karason K, Wigh JP, Dall CH, Gustafsson F, Gullestad L, Nytroen K. Clinical features and determinants of VO2peak in de novo heart transplant recipients. World J Transplant. 2018 Sep 10;8(5):188-197. doi: 10.5500/wjt.v8.i5.188. PMID 30211027
- [Derived] Rafique M, Solberg OG, Gullestad L, Bendz B, Murbraech K, Nytroen K, Rolid K, Lunde K. Effects of high-intensity interval training on cardiac remodelling, function and coronary microcirculation in de novo heart transplant patients: a substudy of the HITTS randomised controlled trial. BMJ Open Sport Exerc Med. 2023 Jul 9;9(3):e001331. doi: 10.1136/bmjsem-2022-001331. eCollection 2023. PMID 37440977
- [Derived] Rolid K, Andreassen AK, Yardley M, Gude E, Bjorkelund E, Authen AR, Grov I, Pettersen KI, Dall CH, Karason K, Broch K, Gullestad L, Nytroen K. High-intensity interval training and health-related quality of life in de novo heart transplant recipients - results from a randomized controlled trial. Health Qual Life Outcomes. 2020 Aug 17;18(1):283. doi: 10.1186/s12955-020-01536-4. PMID 32807179
- [Derived] Nytroen K, Rolid K, Yardley M, Gullestad L. Effect of high-intensity interval training in young heart transplant recipients: results from two randomized controlled trials. BMC Sports Sci Med Rehabil. 2020 Jun 4;12:35. doi: 10.1186/s13102-020-00180-1. eCollection 2020. PMID 32518655
- [Derived] Rolid K, Andreassen AK, Yardley M, Gude E, Bjorkelund E, Authen AR, Grov I, Broch K, Gullestad L, Nytroen K. Long-term effects of high-intensity training vs moderate intensity training in heart transplant recipients: A 3-year follow-up study of the randomized-controlled HITTS study. Am J Transplant. 2020 Dec;20(12):3538-3549. doi: 10.1111/ajt.16087. Epub 2020 Jun 28. PMID 32484261
- [Derived] Nytroen K, Rolid K, Andreassen AK, Yardley M, Gude E, Dahle DO, Bjorkelund E, Relbo Authen A, Grov I, Philip Wigh J, Have Dall C, Gustafsson F, Karason K, Gullestad L. Effect of High-Intensity Interval Training in De Novo Heart Transplant Recipients in Scandinavia. Circulation. 2019 May 7;139(19):2198-2211. doi: 10.1161/CIRCULATIONAHA.118.036747. PMID 30773030